CLINICAL TRIAL: NCT04291859
Title: Interventional, Open-label, Exploratory Study, Investigating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Lu AF28996 in Patients With Parkinson's Disease
Brief Title: Lu AF28996 in Participants With Parkinson's Disease (PD)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18252A; 2019-001280-77 (EudraCT Number)
Record Dates: First submitted 2020-02-28; First posted 2020-03-02 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lu AF28996 (Experimental): Participants in Part A will receive ascending oral doses of Lu AF28996 OD for 14 days in all OD cohorts, followed by down-titration as per Investigator's judgement. For the BID Cohort A1, participants will receive Lu AF28996 BID for 24 days, followed by down-titration as per Investigator's judgement. For the BID Cohort A2, participants will receive Lu AF28996 BID for 39 days, followed by down-titration as per Investigator's judgement.
  Participants in Part B (Cohorts B1, B2, and B3) will receive Lu AF28996 BID for 41 days, followed by down-titration as per Investigator's judgement
  Interventions: Drug: Lu AF28996

INTERVENTIONS:
Drug: Lu AF28996 — capsule, orally, doses and dose escalation scheme will be decided upon at dosing conferences

SUMMARY:
The purpose of this study is to investigate the safety of Lu AF28996, how well it is tolerated and what the body does to the drug in participants with Parkinson's disease.

DETAILED DESCRIPTION:
The study consists of different parts. Part A of the study will consist of once daily (OD) cohorts (OD Cohort 1 to 3), as well as twice daily (BID) cohorts (BID Cohorts A1 and A2). Part B will consist of 3 cohorts (Cohorts B1, B2, and B3) whereby participants will be administered Lu AF28996 BID.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with idiopathic PD (consistent with the UK PD Society Brain Bank Criteria for the Diagnosis of PD), with not more than 1 first-degree relative who has PD.
* Participants must have a Modified Hoehn and Yahr score ≤4 in the OFF state and ≤3 in the ON state, and a Mini Mental State Examination score >25.
* The OFF/ON amplitude on the MDS-UPDRS Part III at screening must be minimum 30% difference.
* Participants must experience recognizable and predictable motor fluctuations (with at least 1.5 hours of OFF periods in the awake time, including predictable morning OFF episodes), causing clinically significant disability during the 7-week Screening Period, as evaluated by the investigator. This will be documented using a participant ON/OFF state registration over 3 consecutive days prior to enrolment.
* Allowed concomitant medication for PD during the study includes levodopa, monoamine oxidase B inhibitors, COMT inhibitors, anticholinergics, and amantadine. Dopamine agonists are not allowed and should be discontinued ≥4 weeks prior to dosing with Lu AF28996 and until the end of the study.
* Participants diagnosed with idiopathic PD (consistent with the UK PD Society Brain Bank Criteria for the Diagnosis of PD), with not more than 1 first-degree relative who has PD.
* Participants must have a Modified Hoehn and Yahr score ≥2 to ≤4 in the OFF state and ≤3 in the ON state, a MDS-UPDRS Part IV, 4.5 score of 1 or 2, and a MDS-UPDRS Part IV, 4.2 score ≥2 (at least mild functional impact), and a Mini Mental State Examination score >25 at the Screening Visit.
* Participants must currently have a good response to levodopa and be receiving a stable dose of levodopa (≥3 doses per day of levodopa/dopa decarboxylase inhibitor therapy or ≥3 doses per day of levodopa Extended-Release Capsules and LEDD between 400 and 1600, inclusive) for at least 4 weeks prior to screening.
* Participants must experience recognizable and predictable motor fluctuations (with ≥3 hours of OFF periods in the awake time, including predictable morning OFF episodes), causing clinically significant disability during 3 months prior to enrolment, as evaluated by the investigator. The criteria will be documented using Hauser Diary over 3 consecutive days prior to enrolment.
* Participants must experience ≥1 hour daily ON time with troublesome dyskinesia (TD) in the awake time (TD/24 hours while awake) during the last 3 months prior to enrolment as evaluated by the investigator. The criteria will be documented using the Hauser Diary over 3 consecutive days prior to enrolment.
* Allowed concomitant medication for PD during the study includes levodopa, dopamine agonists, if allowed daily dose, monoamine oxidase B inhibitors, COMT inhibitors, anticholinergics, and amantadine.

Exclusion Criteria:

* The participant has or had one or more of the following conditions that are considered clinically relevant in the context of the study; other neurological disorder, psychiatric disorder, seizure disorder or encephalopathy, respiratory disease, hepatic impairment or renal insufficiency, metabolic disorder, endocrinological disorder, haematological disorder, infectious disorder, any clinically significant immunological condition, or a history of narrow-angle glaucoma.
* Participant has been treated with apomorphine (pen/pump), and/or inhaled levodopa and/or levodopa/carbidopa intestinal gel (LCIG),and/or subcutaneous foslevodopa/foscarbidopa within 6 weeks prior to the Baseline Visit.
* Participants formerly treated with oral or transdermal dopamine agonists must have discontinued 4 weeks prior to screening.
* Participant has a history of Dopamine Agonist Withdrawal Syndrome (DAWS) when dopamine agonists were previously discontinued or reduced.

Other inclusion and exclusion criteria may apply.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events | From Baseline to 5.5 Months
  Safety and tolerability based on the safety assessments (clinical safety laboratory tests, vital signs, weight, ECG parameters and physical examination)
Cmax of Lu AF28996 | 0 (predose) to 24 hours postdose on Day 1 to Day 47
  Maximum observed plasma concentration of Lu AF28996
Tmax of Lu AF28996 | 0 (predose) to 24 hours postdose on Day 1 to Day 47
  Nominal Time Corresponding to the Occurrence of Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (15):
- United States (9):
  - CenExel Los Alamitos, Los Alamitos, California
  - Georgetown University, Washington D.C., District of Columbia
  - Velocity, Hallandale, Florida
  - Parkinson's Disease Treatment Center of SW FL, Port Charlotte, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - QUEST Research Institute, Farmington Hills, Michigan
  - Neurology Consultants of Nebraska, Omaha, Nebraska
  - Inland Nortwest Research, Spokane, Washington
- Caen Normandy University, Caen, Basse-Normandie, France
- Curiositas-ad-sanum, Hamburg, Germany
- QPS Netherlands BV, Leeuwarden, Netherlands
- Spain (3):
  - Hospital Vall d´Hebron, Barcelona
  - Hosp. General Catalunya, Mira-Sol
  - Virgen Del Roccio, Seville